CLINICAL TRIAL: NCT04773691
Title: Effectiveness of High-frequency rTMS in Reducing Alcohol Consumption in Non-abstinent Patients With an Alcohol Use Disorder: A Multicentre Randomised Controlled Study
Brief Title: Effectiveness of High-frequency rTMS in Reducing Alcohol Consumption in Non-abstinent Patients With an Alcohol Use Disorder
Acronym: ALCOSTIM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TROJAK PHRCI 2014
Record Dates: First submitted 2021-02-24; First posted 2021-02-26 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Alcoholism; rTMS Stimulation
MeSH Terms: conditions — Alcoholism | interventions — Surveys and Questionnaires; Breath Tests

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- test group (Experimental)
  Interventions: Device: Active rTMS; Other: Questionnaires; Device: Breathalyzer
- control group (Placebo Comparator)
  Interventions: Device: Placebo rTMS; Other: Questionnaires; Device: Breathalyzer

INTERVENTIONS:
Device: Active rTMS — Two rTMS stimulation sessions spaced 15 minutes apart are delivered daily for 5 consecutive days.
  A total of 10 sessions. Stimulation parameters: 10 Hz, 1000 pulses per session, 110% of SM, cortical target: right DLPFC
  Arms: test group
Device: Placebo rTMS — Two rTMS stimulation sessions spaced 15 minutes apart are delivered daily for 5 consecutive days.
  A total of 10 sessions. Stimulation parameters: delivering a non-significant current at the beginning and end of the stimulation, simulating active stimulation.
  Arms: control group
Other: Questionnaires — questionnaires for craving assessment: EVA, OCDS, CGI and ADS and signs of physical withdrawal by CIWA
Device: Breathalyzer — estimation of blood alcohol level

SUMMARY:
The fight against alcoholism is a public health priority. Around 15 million Europeans and 10 million North Americans are alcohol dependent. Worldwide, 1 death out of 25 is thought to be attributed to alcohol. In France, the latest published data on alcohol-related mortality indicates that there were 49,000 alcohol-related deaths in 2009. Alcohol is thought to be the leading cause of hospitalisation for French people, and its social cost is estimated at 37.4 billion euros.

However, few patients with an alcohol use disorder are treated: less than 8% in Europe and less than 10.5% in the USA receive appropriate treatment for their alcohol problem. This low rate of treatment is mainly due to the fact that these patients are not ready to stop drinking. They are therefore not attracted by the goal of abstinence that is required by most current therapies and drug treatments. The arrival of new treatments aimed at reducing consumption (rather than abstinence) should make treatment more attractive. To date, nalmefen is the only treatment marketed for this indication. Baclofen should be marketed in 2020, but with restrictive prescription criteria.

In this new strategy to reduce consumption, brain stimulation could play a predominant role as an alternative or complementary therapy. Indeed, functional brain imaging techniques have made it possible to visualise the cortical regions involved in craving, in particular the dorsolateral prefrontal cortex (DLPFC). Craving, i.e. the irrepressible desire to consume, is often at the origin of consumption and relapse. Stimulation of the dorsolateral prefrontal cortex with non-invasive cerebral stimulation techniques, such as repeated transcranial magnetic stimulation (rTMS), has provided encouraging results for the reduction of cravings in all addictive behaviours (alcohol, tobacco, cocaine, food). Furthermore, stimulation of the DLPFC seems to modulate decision-making processes: it may thus reduce impulsivity and strengthen inhibitory control, leading to a reduction in substance use.

The hypothesis to be tested is that repeated transcranial magnetic stimulation allows a reduction in alcohol consumption in patients with an alcohol use disorder.

ELIGIBILITY:
Inclusion Criteria:

* a person who has given his or her free, written and informed consent
* adult patient
* patient with mild to severe alcohol use disorder according to DSM-5 criteria
* voluntary patient to reduce alcohol consumption
* patient who has already made at least one attempt at alcohol withdrawal (failure or relapse), or at reducing consumption

Exclusion Criteria:

* person who is not affiliated to or not a beneficiary of national health insurance
* person subject to a legal protection measure (curatorship, guardianship)
* person subject to a legal safeguard measure
* pregnant, parturient or breastfeeding women
* adult unable to express consent
* patient of childbearing age with a positive pregnancy test at inclusion
* patient with an exhaled alcohol level > 0 milligrams/litre inclusive
* patient with heavy alcohol consumption < 6 days in the 4 weeks prior to inclusion (European Medicine Agency, 2010; one day with alcohol consumption of 60g or more for men and 40g for women)
* patient with an average alcohol consumption below the WHO average risk level in the 4 weeks prior to inclusion (WHO, 2000, less than or equal to 40g/day for men and 40g for women)
* patient being abstinent more than 5 days before inclusion
* patient with a CIWA (Clinical Institute Withdrawal Evaluation: assessment of the severity of alcohol withdrawal) score greater than or equal to 10 at inclusion
* Patient with concomitant treatment with disulfiram, acamprosate, topiramate, baclofen, naltrexone, and nalmefen (< 1 month)
* Patient with a history or presence of pre-delirium tremens or delirium tremens
* Patient with a substance use disorder (DSM-5 criteria) with psychoactive substances other than tobacco and alcohol.
* Patient with acute psychiatric disorders requiring hospitalization and/or immediate adjustment of psychotropic medication
* Patient with severe depression, defined by a score of 24 or more on the Hamilton Depression Scale (HAM-D).
* Patient who has had a recent change (< 1 month) in the prescription of psychotropic treatment
* Patient with severe and/or chronic psychiatric disorders, including schizophrenia, paranoia and bipolar disorders type I and II
* Patient with severe heart, kidney, liver or lung failure or other condition that the doctor believes could compromise the patient's participation in the study.
* Patient with a contraindication to the practice of rTMS; personal history of seizure, pacemaker, neurosurgical clips, carotid or aortic clips, heart valves, hearing aid, ventricular bypass valve, sutures with wires or staples, foreign bodies in the eye, shrapnel, other prosthesis or cephalic ferromagnetic material.
* Patient simultaneously participating in another therapeutic trial
* Patient employed by the investigator or trial site
* Patient who, according to the investigator, is unable to complete a consumption diary and follow up visits for 6 months
* Patient refusing to sign the "safety contract "* specific to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
total alcohol consumption (g/d) | through study completion, an average of 1 month
  total alcohol consumption (g/d), measured by average daily consumption
number of days of high consumption | through study completion, an average of 1 month
  reduction in the number of days of high consumption (≥ 60 g/d for men, ≥ 40 g/d for women)

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Petit B, Soudry-Faure A, Jeanjean L, Foucher J, Lalanne L, Carpentier M, Jonval L, Allard C, Ravier M, Mohamed AB, Meille V, Trojak B. Efficacy of repetitive transcranial magnetic stimulation (rTMS) for reducing consumption in patients with alcohol use disorders (ALCOSTIM): study protocol for a randomized controlled trial. Trials. 2022 Jan 12;23(1):33. doi: 10.1186/s13063-021-05940-z. PMID 35022086